CLINICAL TRIAL: NCT02699944
Title: Optimization of Cardiac Resynchronization Therapy Using an ECG Vest
Brief Title: Optimization of CRT Using an ECG Vest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alan J. Bank, MD (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Alan J. Bank, MD, Medical Director of Research, Allina Health System
Organization: Allina Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 767654-1
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRT sub-optimal responder (Experimental): Subjects who have had CRT for at least 6 months and who have not responded as well as they could, in their cardiologists opinion. Subjects' ejection fraction are still <50% despite CRT. A ECG Vest Optimization protocol will be utilized as one aspect to determine the best CRT programming for each individual subject.
  Interventions: Device: ECG Vest Optimization

INTERVENTIONS:
Device: ECG Vest Optimization — As part of a standard and clinically indicated CRT optimization procedure utilize an ECG Vest as one modality for collecting information to determine best device programming.

SUMMARY:
Despite advancements in implant technology and various techniques of optimization, there is still around 30% non-responder rate to cardiac resynchronization therapy (CRT). This study will assess the potential benefit of a body surface mapping technology to optimize CRT devices in the chronic sub-optimal responder setting.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is one of the most important advances in the treatment of patients with heart failure (HF). This therapy, also known as biventricular pacing, utilizes pacemaker leads to synchronize the contraction of the walls within the left ventricle (LV) and the contraction of the left and right ventricles. Many randomized trials have conclusively demonstrated that CRT improves symptoms, LV structure and function, hospitalization rates, and survival in appropriately selected HF patients. Nonetheless, approximately 30% of CRT patients will be "non-responders" because they will not demonstrate the expected clinical and/or echocardiographic improvement following therapy. A critical component of assessing CRT efficacy during the optimization clinic will be the use of a novel method of body surface electrocardiographic mapping under development by Medtronic, called the ECG Vest. In this proposal, we describe a research study to assess the potential benefit of using the ECG Vest as part of a CRT optimization strategy on clinical and echocardiographic outcomes (heart size and function) of patients receiving standard clinical care in the UHVC CRT Optimization Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients (or their legal guardian) must be willing to provide Informed Consent and a data privacy (HIPPA) authorization
* Patient is or will be followed clinically in the UHVC CRT Optimization Clinic
* Patient has been implanted with a CRT device for at least 6 months
* Patient received an echocardiogram prior to CRT implant
* Patients must be ≥ 18 years of age

Exclusion Criteria:

* Patient's EF is currently ≥ 50%
* Patients who are pregnant
* Patient has unhealed / open wounds on the torso and/or has a history of severe allergic reactions from ECG gel / electrode glue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular end-systolic volume | 6 months after optimization

SECONDARY OUTCOMES:
Determine the degree to which echocardiographic measures of LV function correlate with ECG Vest measures | 6 months after optimization

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Bank, MD, Principal Investigator — Medical Director of Research
Locations (1):
- United Heart & Vascular Clinic, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No